CLINICAL TRIAL: NCT06365151
Title: Effectiveness of an Algorithm for Approaching Temporomandibular Disorders With Osteopathic Manual Therapy in Patients With Fibromyalgia
Brief Title: An Algorithm for Approaching Temporomandibular Disorders With Osteopathic Manual Therapy in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Llanos de la Iglesia, Principal investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMDs fibromyalgia
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia; Temporomandibular Disorder
Keywords: temporomandibular joint disorders; fibromyalgia; Osteopathic medicine; chronic pain; musculoskeletal manipulations
MeSH Terms: conditions — Fibromyalgia; Temporomandibular Joint Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): treatment will be carried out following a previously validated approach algorithm.
  Articulatory techniques, soft tissue mobilization techniques, trigger point inhibition, etc. will be used.
  Interventions: Other: Osteopathic manual therapy
- sham (Sham Comparator): A sham treatment will be performed following a previously validated approach algorithm.
  techniques will be simulated in such a way that they will have no therapeutic effect.
  Interventions: Other: Sham osteopathic manual therapy

INTERVENTIONS:
Other: Osteopathic manual therapy — osteopathic manual treatment aimed at improving the function and pain of the temporomandibular joint.
  Arms: experimental
Other: Sham osteopathic manual therapy — a sham osteopathic manual treatment without therapeutic effect
  Arms: sham

SUMMARY:
Nowadays, fibromyalgia is the rheumatic disorder with the highest levels of deterioration in quality of life. Among the comorbidities it presents, one of the most frequent is temporomandibular disorders. A randomized clinical study will be conducted to evaluate the effectiveness of an osteopathic manual therapy approach algorithm in a group of patients with fibromyalgia and temporomandibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed as suffering from fibromyalgia,
* present moderate pain or dysfunction of more than 3 months' duration in the temporomandibular joint,
* be over 18 years old,
* understand Spanish and/or Catalan correctly,
* and read and accept the informed consent form

Exclusion Criteria:

* history of trauma or recent surgery to the head, face or neck;
* systemic, rheumatic or central nervous system diseases;
* diagnosis of malignant tumors or cancer in the orofacial region;
* participate in other studies at the same time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
catastrophizing | From enrollment to the end of treatment at 6 weeks
  The Pain Catastrophizing scale (PCS), evaluates the degree og catastrophic thinking gdue to pain.It is a 13-item scale, with a total range from 0 to 52. Higher scores are associated with a greater degree of pain catastrophizing.
functional limitation | From enrollment to the end of treatment at 6 weeks
  evaluated with tue short version of the Jaw functional limitation scale (JFLS-8). Evaluates the functional status of the masticatory system. Questionnaire with 8 items, each with a scale from 0 to 10. A higher score suggests a greater limitation.
functional status, disability and pain | From enrollment to the end of treatment at 6 weeks
  collected in the craniofacial pain and disability inventory (CFPDI). Self administered questionnaire of 21 items. Each item is scored on a Likert scale from 0 to 3.
pain and tinnitus | From enrollment to the end of treatment at 6 weeks
  evaluated with a visual analog scale (VAS). Scale from 0 to 10, where 0 indicates no pain and 10 the worst pain imaginable.
myofascial trigger points | From enrollment to 4 weeks
  presence of a palpable tight band, presence of a hyperirritable tenderpoint within te tight band, local twitch response elicited by acute palpation of the tight band, and presence refered pain in response ot trigger point compression.
Range of motion | From enrollment to 4 weeks
  measurements taken with a ruler: maximum opening, maximun active opening without pain and lateralization.

CONTACTS AND LOCATIONS:
Overall Officials: Llanos de la Iglesia, Principal Investigator — Departament de infermeria i fisioterapia. universitat de Lleida
Locations (1):
- Osteopatia i Fisioteràpia Cornellà, Cornellà de Llobregat, Barcelona, Spain